CLINICAL TRIAL: NCT02276170
Title: Pharmacology of Aminophylline for Acute Kidney Injury in Neonates
Acronym: PAANS
Status: Terminated | Type: Observational
Why Stopped: insufficient rate of accrual
Sponsor: Stanford University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Adam R Frymoyer, Clinical Assistant Professor, Stanford University
Other Study IDs: 29957
Record Dates: First submitted 2014-10-21; First posted 2014-10-28 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Aminophylline per standard of care

SUMMARY:
Acute kidney injury (AKI) in critically ill neonates is common and associated with significant morbidity and mortality. No targeted therapeutic treatment strategies have been established for AKI in neonates. Within a clinical pharmacokinetic and pharmacodynamic conceptual framework, this project will examine the medication aminophylline as a potential treatment approach for AKI.

ELIGIBILITY:
Inclusion Criteria:

* Neonate < 3 months post natal age
* Diagnosed with acute kidney injury (AKI)
* Receiving aminophylline for AKI treatment as per local standard of care.

Exclusion Criteria:

* Presence of anatomical renal anomaly based on postnatal evaluation of the patient (hydronephrosis, multicystic kidney, renal agenesis, renal dysplasia, polycystic kidney, or obstructive uropathy)
* Patient on renal replacement therapy
* Major genetic abnormalities (trisomy 13, 18 or 21).

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates with AKI admitted in the NICU who receive aminophylline.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Drug concentrations of theophylline | Day 1 or 2 and Day 3,4, or 5

SECONDARY OUTCOMES:
Change in renal Near-infrared spectroscopy (NIRS) | Day 1,2,3,4
Change in urine output | Day 1,2,3,4
Number of participants with adverse events | 5 days
Change in urine biomarker levels | Day 1,2,3,4,5
Change in serum creatinine level | Day 1,2,3,4,5

CONTACTS AND LOCATIONS:
Overall Officials: Adam Frymoyer, MD, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital Stanford, Palo Alto, California, United States

REFERENCES:
- [Background] Stapleton FB, Jones DP, Green RS. Acute renal failure in neonates: incidence, etiology and outcome. Pediatr Nephrol. 1987 Jul;1(3):314-20. doi: 10.1007/BF00849230. PMID 3153295
- [Background] Agras PI, Tarcan A, Baskin E, Cengiz N, Gurakan B, Saatci U. Acute renal failure in the neonatal period. Ren Fail. 2004 May;26(3):305-9. doi: 10.1081/jdi-200026749. PMID 15354981
- [Background] Koralkar R, Ambalavanan N, Levitan EB, McGwin G, Goldstein S, Askenazi D. Acute kidney injury reduces survival in very low birth weight infants. Pediatr Res. 2011 Apr;69(4):354-8. doi: 10.1203/PDR.0b013e31820b95ca. PMID 21178824
- [Background] Askenazi DJ, Ambalavanan N, Goldstein SL. Acute kidney injury in critically ill newborns: what do we know? What do we need to learn? Pediatr Nephrol. 2009 Feb;24(2):265-74. doi: 10.1007/s00467-008-1060-2. Epub 2008 Dec 10. PMID 19082634
- [Background] Andreoli SP. Acute kidney injury in children. Pediatr Nephrol. 2009 Feb;24(2):253-63. doi: 10.1007/s00467-008-1074-9. Epub 2008 Dec 13. PMID 19083019
- [Background] Mishra J, Dent C, Tarabishi R, Mitsnefes MM, Ma Q, Kelly C, Ruff SM, Zahedi K, Shao M, Bean J, Mori K, Barasch J, Devarajan P. Neutrophil gelatinase-associated lipocalin (NGAL) as a biomarker for acute renal injury after cardiac surgery. Lancet. 2005 Apr 2-8;365(9466):1231-8. doi: 10.1016/S0140-6736(05)74811-X. PMID 15811456
- [Background] Bennett M, Dent CL, Ma Q, Dastrala S, Grenier F, Workman R, Syed H, Ali S, Barasch J, Devarajan P. Urine NGAL predicts severity of acute kidney injury after cardiac surgery: a prospective study. Clin J Am Soc Nephrol. 2008 May;3(3):665-73. doi: 10.2215/CJN.04010907. Epub 2008 Mar 12. PMID 18337554
- [Background] Askenazi DJ, Griffin R, McGwin G, Carlo W, Ambalavanan N. Acute kidney injury is independently associated with mortality in very low birthweight infants: a matched case-control analysis. Pediatr Nephrol. 2009 May;24(5):991-7. doi: 10.1007/s00467-009-1133-x. Epub 2009 Feb 24. PMID 19238451
- [Background] Mangione F, Calcaterra V, Esposito C, Dal Canton A. Renal blood flow redistribution during acute kidney injury. Am J Kidney Dis. 2010 Oct;56(4):785-7. doi: 10.1053/j.ajkd.2010.03.035. Epub 2010 Jun 26. PMID 20580475
- [Background] Voors AA, Dittrich HC, Massie BM, DeLucca P, Mansoor GA, Metra M, Cotter G, Weatherley BD, Ponikowski P, Teerlink JR, Cleland JG, O'Connor CM, Givertz MM. Effects of the adenosine A1 receptor antagonist rolofylline on renal function in patients with acute heart failure and renal dysfunction: results from PROTECT (Placebo-Controlled Randomized Study of the Selective Adenosine A1 Receptor Antagonist Rolofylline for Patients Hospitalized with Acute Decompensated Heart Failure and Volume Overload to Assess Treatment Effect on Congestion and Renal Function). J Am Coll Cardiol. 2011 May 10;57(19):1899-907. doi: 10.1016/j.jacc.2010.11.057. PMID 21545947
- [Background] Lee HT, Xu H, Nasr SH, Schnermann J, Emala CW. A1 adenosine receptor knockout mice exhibit increased renal injury following ischemia and reperfusion. Am J Physiol Renal Physiol. 2004 Feb;286(2):F298-306. doi: 10.1152/ajprenal.00185.2003. Epub 2003 Nov 4. PMID 14600029
- [Background] Jenik AG, Ceriani Cernadas JM, Gorenstein A, Ramirez JA, Vain N, Armadans M, Ferraris JR. A randomized, double-blind, placebo-controlled trial of the effects of prophylactic theophylline on renal function in term neonates with perinatal asphyxia. Pediatrics. 2000 Apr;105(4):E45. doi: 10.1542/peds.105.4.e45. PMID 10742366
- [Background] Bakr AF. Prophylactic theophylline to prevent renal dysfunction in newborns exposed to perinatal asphyxia--a study in a developing country. Pediatr Nephrol. 2005 Sep;20(9):1249-52. doi: 10.1007/s00467-005-1980-z. Epub 2005 Jun 10. PMID 15947981
- [Background] Bhat MA, Shah ZA, Makhdoomi MS, Mufti MH. Theophylline for renal function in term neonates with perinatal asphyxia: a randomized, placebo-controlled trial. J Pediatr. 2006 Aug;149(2):180-4. doi: 10.1016/j.jpeds.2006.03.053. PMID 16887430